CLINICAL TRIAL: NCT03458455
Title: Improved Therapy Response Assessment in Metastatic Brain Tumors
Acronym: TREATMENT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Hospital of Southern Norway Trust (Other); Ostfold Hospital Trust (Other); St. Olavs Hospital (Other); Massachusetts General Hospital (Other); Dana-Farber Cancer Institute (Other); University Medical Center Groningen (Other); University of Texas Southwestern Medical Center (Other); South-Eastern Norway Regional Health Authority (Other); Norwegian Cancer Society (Other)
Responsible Party: Principal Investigator, Kyrre Eeg Emblem, Principal Investigator, Oslo University Hospital
Other Study IDs: 2013/1033 LOOPS
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Brain Metastases
Keywords: TREATMENT; Vessel Architectural Imaging; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Imaging; Radiosurgery; Ipilimumab; Nivolumab; pembrolizumab; Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (5):
- A: Patients with brain metastases from non-small cell lung cancer receiving stereotactic radiosurgery to selected lesions
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Radiation: Stereotactic Radiosurgery
- B: Patients with brain metastases from malignant melanoma receiving stereotactic radiosurgery to selected lesions
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Radiation: Stereotactic Radiosurgery
- C: Patients with brain metastases from non-small cell lung cancer receiving stereotactic radiosurgery to selected lesions + nivolumab or pembrolizumab
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Radiation: Stereotactic Radiosurgery; Drug: Ipilimumab, nivolumab or pembrolizumab
- D: Patients with brain metastases from malignant melanoma receiving stereotactic radiosurgery to selected lesions + ipilimumab, nivolumab or pembrolizumab
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Radiation: Stereotactic Radiosurgery; Drug: Ipilimumab, nivolumab or pembrolizumab
- E: Patients with brain metastases from non-small cell lung cancer receiving stereotactic radiosurgery to selected lesions + epidermal growth factor receptor (EGFR) inhibitors
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Vessel Architectural Imaging is an MRI-based tumor diagnostic framework providing a powerful tool for non-invasive, in vivo assessment of diagnostic biomarkers relevant for these new therapy forms; microvascular function and tumor oxygenation.
  Other Names: Vessel Architectural Imaging
Radiation: Stereotactic Radiosurgery — A non-surgical radiation therapy used to treat tumors of the brain. It can deliver precisely-targeted radiation in fewer high-dose treatments than traditional therapy, which can help preserve healthy tissue.
Drug: Ipilimumab, nivolumab or pembrolizumab — A type of therapy that uses substances to stimulate the immune system to help the body fight cancer by blocking inhibitory receptors on lymphocytes to overcome immune tolerance.
  Other Names: Immunotherapy
  Groups: C; D

SUMMARY:
TREATMENT is an observational study addressing the need for knowledge and adequate diagnostic biomarkers in the response assessment of patients with brain metastasis. Reliable response assessment will be highly relevant in the coming years given the introduction of next-generation cancer drugs, including immunotherapy. This project uses advanced Magnetic Resonance Imaging (MRI) and Vessel Architecture Imaging (VAI) to better understand the response to traditional stereotactic radiosurgery (SRS) and immunotherapy.

Secondary objectives include:

In patients with brain metastases, use advanced MRI and Vessel Architectural Imaging methods to reveal parameters of traditional, immunotherapeutic, and anti-angiogenic therapy response.

In patients with brain metastases, use advanced MRI and Vessel Architectural Imaging methods to compare results with traditional biomarkers.

Use existing infrastructure at Oslo University Hospital to standardize therapy monitoring.

In patients with brain metastases, use advanced MRI and Vessel Architectural Imaging methods to separate real tumor progression from treatment-induced pseudoprogression or radionecrosis

In patients with brain metastases, use advanced MRI and Vessel Architectural Imaging methods to assess whether anti-angiogenic drugs improve delivery of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically - or - radiographically confirmed metastatic disease from a primary non-small-cell lung cancer - or - metastatic melanoma.
* Participants must have measurable disease in the central nervous system (CNS), defined as at least one lesion that can be accurately measured in at least one dimension as ≥5 mm with MRI - or - compromise more than 30 image voxels on perfusion MRI to ensure adequate parametric statistical assessments. For a perfusion MRI resolution of 1.2x1.2x5mm, this equals a tumor volume of 0.2cubic centimeters (cc).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1 (Karnofsky ≥60%)
* Life expectancy of greater than 6 weeks
* Eligible for stereotactic radiosurgery
* Have normal organ functions per clinical guidelines
* Ability to understand and the willingness to sign a written informed consent document.
* Previously untreated asymptomatic brain metastases - or - progressive brain metastases after systemic therapy or prior local therapy such as radiation or surgery as defined by:

  1. Untreated measurable lesions in patients that have received surgery and/or SRS to one or more other lesions
  2. Residual or progressive lesions after surgery if asymptomatic
  3. Patients who have had prior whole-brain radiation therapy (WBRT) and/or SRS and then whose lesions have progressed are eligible. Lesions treated with SRS may be eligible if there is unequivocal evidence of progression
  4. Progression after prior systemic therapy.

Exclusion Criteria:

* Participants who received major surgery must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a diagnosis of immunodeficiency or hypersensitivity to ipilimumab or any of its excipients (Cohorts C and D).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a known additional malignancy that is progressing or requires active treatment.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Unable to undergo brain MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both men and women of all races and ethnic groups are eligible for this trial.
  Cohort A: Accrual of up to 55 patients with brain metastases from NSCLC may be required in order to achieve 50 evaluable patients.
  Cohort B: Accrual of up to 33 patients with brain metastases from malignant melanomas may be required in order to achieve 30 evaluable patients.
  Cohort C: Accrual of up to 55 patients with brain metastases from malignant melanomas may be required in order to achieve 50 evaluable patients.
  Cohort D: Accrual of up to 33 patients with brain metastases from malignant melanomas may be required in order to achieve 30 evaluable patients.
  Cohort E: Accrual of up to 22 patients with brain metastases from malignant melanomas may be required in order to achieve 20 evaluable patients.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-03-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Response | 18 months
  Radionecrosis, pseudoprogression or tumor progression by Response Assessment in Neuro-Oncology Criteria (RANO) or histology, or radiographic/clinical progression free survival

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Kyrre E Emblem, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Within one year following study end, anonymized data will be uploaded to the appropriate online repositories to promote open access. This anonymized data includes general clinical information deemed non-identifiable (age, weight, gender, diagnosis and any prior treatments), imaging data (MRI with exam intervals only, no dates), corresponding results of any tissue analyses as well as study treatments (with treatment doses and intervals, no dates).

REFERENCES:
- [Background] Gerstner ER, Emblem KE, Sorensen GA. Vascular Magnetic Resonance Imaging in Brain Tumors During Antiangiogenic Therapy--Are We There Yet? Cancer J. 2015 Jul-Aug;21(4):337-42. doi: 10.1097/PPO.0000000000000128. PMID 26222087
- [Background] Emblem KE, Farrar CT, Gerstner ER, Batchelor TT, Borra RJ, Rosen BR, Sorensen AG, Jain RK. Vessel caliber--a potential MRI biomarker of tumour response in clinical trials. Nat Rev Clin Oncol. 2014 Oct;11(10):566-84. doi: 10.1038/nrclinonc.2014.126. Epub 2014 Aug 12. PMID 25113840
- [Background] Emblem KE, Mouridsen K, Bjornerud A, Farrar CT, Jennings D, Borra RJ, Wen PY, Ivy P, Batchelor TT, Rosen BR, Jain RK, Sorensen AG. Vessel architectural imaging identifies cancer patient responders to anti-angiogenic therapy. Nat Med. 2013 Sep;19(9):1178-83. doi: 10.1038/nm.3289. Epub 2013 Aug 18. PMID 23955713
- [Background] Lin NU, Lee EQ, Aoyama H, Barani IJ, Barboriak DP, Baumert BG, Bendszus M, Brown PD, Camidge DR, Chang SM, Dancey J, de Vries EG, Gaspar LE, Harris GJ, Hodi FS, Kalkanis SN, Linskey ME, Macdonald DR, Margolin K, Mehta MP, Schiff D, Soffietti R, Suh JH, van den Bent MJ, Vogelbaum MA, Wen PY; Response Assessment in Neuro-Oncology (RANO) group. Response assessment criteria for brain metastases: proposal from the RANO group. Lancet Oncol. 2015 Jun;16(6):e270-8. doi: 10.1016/S1470-2045(15)70057-4. Epub 2015 May 27. PMID 26065612
- [Background] Lin NU, Wefel JS, Lee EQ, Schiff D, van den Bent MJ, Soffietti R, Suh JH, Vogelbaum MA, Mehta MP, Dancey J, Linskey ME, Camidge DR, Aoyama H, Brown PD, Chang SM, Kalkanis SN, Barani IJ, Baumert BG, Gaspar LE, Hodi FS, Macdonald DR, Wen PY; Response Assessment in Neuro-Oncology (RANO) group. Challenges relating to solid tumour brain metastases in clinical trials, part 2: neurocognitive, neurological, and quality-of-life outcomes. A report from the RANO group. Lancet Oncol. 2013 Sep;14(10):e407-16. doi: 10.1016/S1470-2045(13)70308-5. PMID 23993385
- [Background] Lin NU, Lee EQ, Aoyama H, Barani IJ, Baumert BG, Brown PD, Camidge DR, Chang SM, Dancey J, Gaspar LE, Harris GJ, Hodi FS, Kalkanis SN, Lamborn KR, Linskey ME, Macdonald DR, Margolin K, Mehta MP, Schiff D, Soffietti R, Suh JH, van den Bent MJ, Vogelbaum MA, Wefel JS, Wen PY; Response Assessment in Neuro-Oncology (RANO) group. Challenges relating to solid tumour brain metastases in clinical trials, part 1: patient population, response, and progression. A report from the RANO group. Lancet Oncol. 2013 Sep;14(10):e396-406. doi: 10.1016/S1470-2045(13)70311-5. PMID 23993384
- [Result] Digernes I, Bjornerud A, Vatnehol SAS, Lovland G, Courivaud F, Vik-Mo E, Meling TR, Emblem KE. A theoretical framework for determining cerebral vascular function and heterogeneity from dynamic susceptibility contrast MRI. J Cereb Blood Flow Metab. 2017 Jun;37(6):2237-2248. doi: 10.1177/0271678X17694187. Epub 2017 Jan 1. PMID 28273722
- [Result] Angeli S, Emblem KE, Due-Tonnessen P, Stylianopoulos T. Towards patient-specific modeling of brain tumor growth and formation of secondary nodes guided by DTI-MRI. Neuroimage Clin. 2018 Aug 31;20:664-673. doi: 10.1016/j.nicl.2018.08.032. eCollection 2018. PMID 30211003
- [Result] Nilsen LB, Digernes I, Grovik E, Saxhaug C, Latysheva A, Geier O, Breivik B, Saetre DO, Jacobsen KD, Helland A, Emblem KE. Responses in the diffusivity and vascular function of the irradiated normal brain are seen up until 18 months following SRS of brain metastases. Neurooncol Adv. 2020 Feb 28;2(1):vdaa028. doi: 10.1093/noajnl/vdaa028. eCollection 2020 Jan-Dec. PMID 32642687
- [Result] Seano G, Nia HT, Emblem KE, Datta M, Ren J, Krishnan S, Kloepper J, Pinho MC, Ho WW, Ghosh M, Askoxylakis V, Ferraro GB, Riedemann L, Gerstner ER, Batchelor TT, Wen PY, Lin NU, Grodzinsky AJ, Fukumura D, Huang P, Baish JW, Padera TP, Munn LL, Jain RK. Solid stress in brain tumours causes neuronal loss and neurological dysfunction and can be reversed by lithium. Nat Biomed Eng. 2019 Mar;3(3):230-245. doi: 10.1038/s41551-018-0334-7. Epub 2019 Jan 7. PMID 30948807
- [Result] Digernes I, Grovik E, Nilsen LB, Saxhaug C, Geier O, Reitan E, Saetre DO, Breivik B, Reese T, Jacobsen KD, Helland A, Emblem KE. Brain metastases with poor vascular function are susceptible to pseudoprogression after stereotactic radiation surgery. Adv Radiat Oncol. 2018 May 17;3(4):559-567. doi: 10.1016/j.adro.2018.05.005. eCollection 2018 Oct-Dec. PMID 30370356
- See also: Brain metastases with poor vascular function are susceptible to pseudoprogression after stereotactic radiation surgery — https://linkinghub.elsevier.com/retrieve/pii/S2452109418300836